CLINICAL TRIAL: NCT05137743
Title: Pilot Test of Apnea and Insomnia Relief for Veterans With Gulf War Illness
Acronym: GWAIR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); CDMRP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-33521; CDMRP - GW200046 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gulf War Illness

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with participants assigned to one of two treatment groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: The study statistician who will analyze outcome data will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apnea and Insomnia Relief (AIR) (Experimental): This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. The main components of the AIR protocol are (a) psychoeducation, (b) motivational interviewing, (c) PAP adherence strategies, and (d) cognitive behavioral therapy for insomnia (CBT-I).
  Interventions: Behavioral: Apnea and Insomnia Relief (AIR)
- Sleep Education (SE) (Active Comparator): This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. Topics covered include the sleep cycle, sleep across the lifespan, sleep and the mind, evening activities and the sleep environment, and daytime activities and sleep.
  Interventions: Behavioral: Sleep Education (SE)

INTERVENTIONS:
Behavioral: Apnea and Insomnia Relief (AIR) — This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. The main components of the AIR protocol are (a) psychoeducation, (b) motivational interviewing, (c) PAP adherence strategies, and (d) cognitive behavioral therapy for insomnia.
  Arms: Apnea and Insomnia Relief (AIR)
Behavioral: Sleep Education (SE) — This treatment will be offered over six sessions. All appointments will be conducted via telehealth and will last 60 minutes. Topics covered include the sleep cycle, sleep across the lifespan, sleep and the mind, evening activities and the sleep environment, and daytime activities and sleep.
  Arms: Sleep Education (SE)

SUMMARY:
The purpose of this study is to determine whether a behavioral sleep treatment improves sleep and other Gulf War Illness (GWI) symptoms in Gulf War Veterans with GWI.

DETAILED DESCRIPTION:
This study is a randomized controlled trial of a behavioral sleep treatment to improve sleep and other symptoms of Gulf War Illness (GWI) in Gulf War (GW) Veterans with GWI, sleep apnea, and insomnia. The treatment is delivered via telehealth (video to home) or telephone. The primary outcome for this study is the severity of Gulf War Illness symptom severity. Other outcomes include sleep-related functioning, insomnia symptom severity, and positive airway pressure (PAP) adherence.

ELIGIBILITY:
Inclusion Criteria:

* Male and female GW Veterans between the ages of 48-80
* Deployed to the "Gulf Theater of operations," as defined by 38 CFR 3.317
* Meets the Kansas GWI and Centers for Disease Control and Prevention (CDC) Chronic Multisymptom Illness (CMI) case definitions. The Kansas GWI definition requires cases to endorse multiple or moderate-to-severe chronic symptoms in at least three of six symptom domains. These include: i) fatigue/sleep problems, ii) somatic pain, iii) neurological cognitive, mood symptoms, iv) gastrointestinal symptoms, v) respiratory symptoms, and vi) skin abnormalities. Veterans will be excluded from being considered Kansas GWI cases, for purposes of the proposed trial, if they report being diagnosed by a physician with medical or psychiatric conditions that would account for their symptoms or interfere with their ability to report their symptoms. Veterans with current or past history of PTSD or depression in the past 5 years will not be excluded from participation if they have not been hospitalized for these conditions. The CDC CMI case definition requires cases to endorse symptoms in at least two of three symptom clusters. These include: i) fatigability (e.g., feeling fatigue for 24 hours or more after exertion), ii) mood/cognitive symptoms (e.g., feeling depressed, irritable, worried, tense or anxious; difficulty thinking or concentrating, problems finding words, or problems getting to or staying asleep). iii) musculoskeletal pain.
* Meet the DSM-5 research diagnostic criteria for insomnia disorder. Unlike other GWI symptoms, we will not require the Veteran's insomnia to have begun during the Gulf War or within one year after leaving the Gulf region. This is because some GWI symptoms may cause veterans to adopt behaviors that lead to sleep problems later. Results from our CBT-I trial in Veterans with GWI suggest that improving sleep also improves non-sleep related symptoms such as fatigue, depression, pain, and psychosocial function. Therefore, we hypothesize that even if insomnia was not one of the original GWI symptoms, improving sleep in veterans with GWI will also improve other GWI-related symptoms.
* Diagnosed with obstructive sleep apnea (OSA) by physician based on polysomnography or evidence of OSA based on an Apnea-Hyponea Index (AHI) or respiratory disturbance index (RDI) that is > or = 5 based on home sleep apnea testing.
* Have access to wireless internet connection at home for remote positive airway pressure (PAP) data capture.

Exclusion Criteria:

* Condition(s) that is/are considered exclusionary for the Kansas GWI criteria. For purposes of this trial, this will include medical or psychiatric conditions diagnosed by a physician/psychiatrist that would account for the Veterans' symptoms or interfere with their ability to report their symptoms. Specific exclusionary criteria include medical conditions such as uncontrolled diabetes, heart disease other than hypertension, stroke, lupus, multiple sclerosis, cancer, liver disease, chronic infection, or serious neurological condition (e.g., dementia, brain injury).
* History of any psychiatric disorder with active psychosis or mania in the past 5 years.
* Severe drug or alcohol use disorder within the past 6 months as assessed by the Structured Clinical Interview for DSM-5 (SCID 5). Veterans with moderate drug or alcohol use disorder will be reviewed on a case-by-case basis.
* Prominent suicidal or homicidal ideation.
* Pregnancy, because insomnia will worsen after 8 weeks.
* Restless Legs Syndrome (RLS) or screening indicative of RLS based on Restless legs syndrome screening questionnaire (RLSSQ).
* Current enrollment in another clinical trial.
* Traumatic brain injury (TBI) will not be exclusionary for the proposed study unless it impacts cognition to a degree that the Veteran cannot complete treatment or homework assignments (this will be determined on a case-by-case basis at PI and therapists' discretion).
* Starting or ending psychotherapy for a sleep disorder or mental health diagnosis within the last one month.
* Starting or ending an antidepressant, anxiolytic, or sleep medication with the last one month will be excluded. Veterans currently receiving benzodiazepine or benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, or non-SSRI antidepressant medications such as trazodone will be not be excluded provided that they meet the DSM-5 criteria for insomnia disorder, exhibit evidence of OSA, and will remain on the medication(s) throughout the 6-week treatment period and the 3-month follow-up period.

Ages: 48 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Gulf War Illness Symptom Severity Index | Change from baseline to 1 week post-treatment (after 6 weeks).
  Due to its novelty, complexity, and variability, no single measure of severity addresses all possible presentations of Gulf War Illness (GWI). Therefore, we used the symptom portion of the Kansas Gulf War Military History and Health Questionnaire to query about fatigue/sleep problems, somatic pain, skin abnormalities, gastrointestinal, respiratory, and neurologic/cognitive/mood symptoms, based on the Kansas GWI and CDC CMI case definition. To assess current GWI symptoms, participants will be asked about the absence (0), presence, and severity (1=mild; 2=moderate; 3=severe) of the symptoms over the past 2 weeks instead of over the past 6-months. Score range: 0-87; higher scores = more symptoms and/or more severe symptoms.
Change in Gulf War Illness Symptom Severity Index | Change from baseline to 3 months after treatment ends.
  Due to its novelty, complexity, and variability, no single measure of severity addresses all possible presentations of Gulf War Illness (GWI). Therefore, we used the symptom portion of the Kansas Gulf War Military History and Health Questionnaire to query about fatigue/sleep problems, somatic pain, skin abnormalities, gastrointestinal, respiratory, and neurologic/cognitive/mood symptoms, based on the Kansas GWI and CDC CMI case definition. To assess current GWI symptoms, participants will be asked about the absence (0), presence, and severity (1=mild; 2=moderate; 3=severe) of the symptoms over the past 2 weeks instead of over the past 6-months. Score range: 0-87; higher scores = more symptoms and/or more severe symptoms.
Change in Positive Airway Pressure (PAP) Adherence | Change from baseline to 1 week post-treatment (after 6 weeks).
  PAP adherence will be measured via PAP device data capture. The average hours of PAP use will be measured from session 1 through post-treatment.
Positive Airway Pressure (PAP) Adherence | Change from baseline to 3 months after treatment ends.
  PAP adherence will be measured via PAP device data capture. The average hours of PAP use will be measured for 1 week at the follow-up 3 months after treatment ends.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | Change from baseline to 1 week post-treatment (after 6 weeks).
  This seven-item self-report scale assesses severity of insomnia. Responses to items range from 0 to 4. Total scores range from 0 to 28. Higher scores indicate greater symptom severity.
Insomnia Severity Index (ISI) | Change from baseline to 3 months after treatment ends.
  This seven-item self-report scale assesses severity of insomnia. Responses to items range from 0 to 4. Total scores range from 0 to 28. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Chao, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chao LL, Kanady JC, Crocker N, Straus LD, Hlavin J, Metzler TJ, Maguen S, Neylan TC. Cognitive behavioral therapy for insomnia in veterans with gulf war illness: Results from a randomized controlled trial. Life Sci. 2021 Aug 15;279:119147. doi: 10.1016/j.lfs.2021.119147. Epub 2021 Feb 4. PMID 33549595